CLINICAL TRIAL: NCT07389850
Title: Evaluation of the Evolution of Proprioceptive Reweighting Abilities Following Anterior Cruciate Ligament Reconstruction Surgery - ReproEVO
Brief Title: Evaluation of the Evolution of Proprioceptive Reweighting Abilities Following Anterior Cruciate Ligament Reconstruction Surgery
Acronym: ReproEVO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 29BRC25.0312
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Anterior Cruciate Ligament Rupture With Ligamentoplasty
Keywords: Anterior Cruciate Ligament; Anterior Cruciate Ligament Reconstruction; Central Nervous System; Proprioceptive reweighting; Pivot-contact sport; Plastic patient; Athletes

STUDY DESIGN:
Intervention Model Description: ReproEVO is a multicenter prospective interventional study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Anterior Cruciate Ligament (Experimental): Patients with Anterior Cruciate Ligament (ACL) rupture scheduled for ACL reconstruction surgery
  Interventions: Procedure: ReproEVO intervention

INTERVENTIONS:
Procedure: ReproEVO intervention — After the inclusion visit, each assessment will include an examination of standing balance in two support conditions: hard floor or soft floor and two conditions of vibration of the Achilles tendons or lumbar muscles, performed randomly over five trials for each condition. The subjects stand with their eyes covered by an opaque mask. Vibrators are positioned at both locations and vibrated randomly after a trial without recording to perceive the destabilizing effect induced by the vibration. The data is recorded using a force platform on the floor.
  Subjects will be seated and strapped into a rigid device attached to their leg. The device is connected to a motor that maintains a constant speed. Maximum strength will be measured at two different speeds.
  Finally, at each assessment, the subjects will complete questionnaires about their fear of pain, their assessment of their knee's capabilities, and the activities they engage in.

SUMMARY:
Anterior cruciate ligament (ACL) injury is the most common knee injury among athletes who play contact sports involving pivoting. ACL reconstruction (ACLR) combined with rehabilitation is the standard treatment for ACL tears in athletes, and rehabilitation is one of the keys to success. The overall return to sport rate is 80%, but the return to pre-injury level of sport is only 65% and the return to the same level of competition is only 55%. The recurrence rate is close to 20%.

During rehabilitation and sports practice, proprioceptive information is essential for adjusting the muscle sensorimotor loop and enabling optimal movement.

Athletes can thus be classified as plastic or rigid . Our hypothesis is to show that the proportion of "plastic" patients 9 months post-operative following ACL reconstruction is higher than that found in the same population 3 months post-operative, thus demonstrating the progression of proprioceptive integration abilities after ACL reconstruction surgery.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) injury is the most common knee injury among athletes who play contact sports involving pivoting. ACL reconstruction (ACLR) combined with rehabilitation is the standard treatment for ACL tears in athletes, and rehabilitation is one of the keys to success. The overall return to sport rate is 80%, but the return to pre-injury level of sport is only 65% and the return to the same level of competition is only 55%. The recurrence rate is close to 20%. Although the number of studies on the subject is growing, there is currently no consensus on rehabilitation protocols.

During rehabilitation and sports practice, proprioceptive information is essential for adjusting the muscle sensorimotor loop and enabling optimal movement.

We have demonstrated that athletes and athletes after ACL reconstruction show variability in the integration of proprioceptive information during a complex balance task.

Athletes can thus be classified as plastic (able to vary the source of proprioceptive information depending on conditions) or rigid (unable to do so).

Our hypothesis is to show that the proportion of "plastic" patients 9 months post-operative following ACL reconstruction is higher than that found in the same population 3 months post-operative, thus demonstrating the progression of proprioceptive integration abilities after ACL reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 15 and 40;
* Patients with ACL rupture scheduled for ACL reconstruction surgery;
* Patients able to maintain a stable bipedal standing position without technical assistance and with their eyes closed;
* Consent of the patient, parents, legal guardians, or guardians to the recording (for minor patients) of data for research and publication purposes.

Exclusion Criteria:

* Recent osteoarticular pathology (i.e., less than three months) of the lower limbs, whether traumatic or not, other than ACL rupture;
* Proven disabling neurological pathology;
* Pain in the musculoskeletal system during exercise (excluding the operated knee);
* Fatigue assessed using the Borg scale > 6;
* Skin allergy to an adhesive product.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2028-05-20 (Estimated); Study Completion 2028-05-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of progress in proprioceptive reweighting after knee ligament reconstruction | Baseline, 3 months after surgery and 9 months after surgery
  Difference between the mean proprioceptive reweighting coefficient (RPw) preoperatively and 3 months postoperatively

SECONDARY OUTCOMES:
Assesment of the variation in weighting between before and after the operation | Baseline and 3 months postoperatively
  Difference between the mean proprioceptive reweighting coefficient (RPw) preoperatively and 3 months postoperatively
Assess postural control | Baseline, at 3 months postoperatively and at 9 months postoperatively
  Difference in the size of the shift in the center of pressure in a static standing position, with eyes open and closed
Assess your Anterior Cruciate Ligament - Return to Sport and Injury (ACL-RSI) perception score | Baseline, at 3 months postoperatively and at 9 months postoperatively
  Assess your Anterior Cruciate Ligament - Return to Sport and Injury (ACL-RSI) perception score (0 : Not at all sure; 10: Completely safe) at the inclusion visit (preoperative); at 3 months postoperatively and at 9 months postoperatively
Assess the subjective IKDC activity score | Baseline, at 3 months postoperatively and at 9 months postoperatively
  Assess the subjective IKDC activity score (0: Never; 10: Always) at the inclusion visit (preoperative); at 3 months postoperatively and at 9 months postoperatively.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Brest University Hospital, Brest
  - Montpellier University Hospital, Montpellier
  - Dr. STER Clinic, Saint Clément de Rivière, Saint-Clément-de-Rivière

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.